CLINICAL TRIAL: NCT02364375
Title: Menai Mask Systems - Clinical Study 1
Brief Title: Usability Evaluation of Menai CPAP Masks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MA220115
Record Dates: First submitted 2015-02-01; First posted 2015-02-18 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep; apnea; OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Face (Experimental): Participants will trial the same mask type/variant (full face, nasal, pillows) as the variant they are using as part of their current treatment. Participants in this arm will trial the Menai mask (full face) and Comparison Menai Standard mask (full face) for 7 nights each.
  Interventions: Device: Menai mask (full face); Device: Menai Standard mask (full face)
- Nasal (Experimental): Participants will trial the same mask type/variant (full face, nasal, pillows) as the variant they are using as part of their current treatment. Participants in this arm will trial the Menai mask (nasal) and Comparison Menai Standard mask (nasal) for 7 nights each.
  Interventions: Device: Menai mask (nasal); Device: Menai Standard mask (nasal)
- Pillows (Experimental): Participants will trial the same mask type/variant (full face, nasal, pillows) as the variant they are using as part of their current treatment. Participants in this arm will trial the Menai mask (pillows) and Comparison Menai Standard mask (pillows) for 7 nights each.
  Interventions: Device: Menai mask (pillows); Device: Menai Standard mask (pillows)

INTERVENTIONS:
Device: Menai mask (full face) — Prototype mask system (full face variant) with novel vent and humidification system
  Arms: Full Face
Device: Menai Standard mask (full face) — Prototype mask system (full face variant) with conventional vent and humidification system
  Arms: Full Face
Device: Menai mask (nasal) — Prototype mask system (nasal variant) with novel vent and humidification system
  Arms: Nasal
Device: Menai Standard mask (nasal) — Prototype mask system (nasal variant) with conventional vent and humidification system
  Arms: Nasal
Device: Menai mask (pillows) — Prototype mask system (pillows variant) with conventional vent and humidification system
  Arms: Pillows
Device: Menai Standard mask (pillows) — Prototype mask system (pillows variant) with conventional vent and humidification system
  Arms: Pillows

SUMMARY:
The primary objective of this study is to evaluate the subjective performance of the Menai mask systems (full face, nasal, and pillows variants), compared against Comparison mask systems.

DETAILED DESCRIPTION:
The study will evaluate the subjective seal, comfort, stability, usability, and humidification performance of the prototype mask systems in CPAP established patients. The performance of the prototype Menai mask systems (full face, nasal, and pillows variants) will be subjectively assessed through user questionnaires based on an 11-point Likert scale, and will be compared against Comparison masks.

The prototype masks share the same parts (cushion, frame, headgear), with the difference being that the Menai masks feature a novel vent and humidification system.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to provide written informed consent
* Participants who can read and comprehend written and spoken English
* Participants who are over 18 years of age
* Participants who have been diagnosed with OSA
* Participants who have been established on CPAP for ≥ 6 months
* Participants who are currently using the same mask type/variant as the interventional mask system to be evaluated

Exclusion Criteria:

* Participants who are not able to provide written informed consent
* Participants who are unable to comprehend written and spoken English
* Participants who are pregnant
* Participants who are unsuitable to participate in the study in the opinion of the researcher
* Participants with a pre-existing lung disease or a condition that would predispose them to pneumothorax (e.g. COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection, lung injury)
* Participants who cannot participate for the duration of the trial
* Participants who are established on bi-level support therapy
* Participants who are not currently using the same mask type/variant as the interventional mask system to be evaluated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Usability Performance Evaluation | 2 weeks
  Evaluation of the usability performance (seal, comfort, etc) of the Menai masks, compared to the Comparison Menai Standard masks.

SECONDARY OUTCOMES:
Humidification Performance Evaluation | 2 weeks
  Evaluation of the humidification performance of the Menai masks (passive humidification), compared to the Comparison Menai Standard masks (active humidification).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, BE PhD, Principal Investigator — Graduate School of Biomedical Engineering, University of New South Wales, Sydney Australia and Applied Research, ResMed Ltd Sydney Australia
Locations (1):
- ResMed Sleep Research Centre, Sydney, New South Wales, Australia